CLINICAL TRIAL: NCT07032597
Title: A Multicenter, Evaluator Blinded, Randomized Study to Evaluate the Safety and Effectiveness of HArmonyCa Lidocaine Compared to Restylane® Perlane® Lidocaine for Restoration and/or Creation of Mid-face Volume
Brief Title: A Study to Assess Safety and Effectiveness of HArmonyCa Lidocaine Injectable Gel for Restoration and/or Creation of Mid-Face Volume in Adult Participants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M21-782
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Mid Face Volume Deficit
Keywords: Mid Face Volume Deficit; HArmonyCa Lidocaine; Restylane® Perlane® Lidocaine; Mid-Face China

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HArmonyCa Lidocaine (Experimental): Participants will receive HArmonyCa Lidocaine on Day 1 with optional touch-up treatment on Day 31.
  Interventions: Device: HArmonyCa Lidocaine Injectable Gel
- Restylane® Perlane® Lidocaine (Active Comparator): Participants will receive Perlane on Day 1 with optional touch-up treatment on Day 31.
  Interventions: Device: Restylane® Perlane® Lidocaine

INTERVENTIONS:
Device: HArmonyCa Lidocaine Injectable Gel — Subdermal or Deep Dermal or Supraperiosteal Injection
  Arms: HArmonyCa Lidocaine
Device: Restylane® Perlane® Lidocaine — Subcutaneous to Supraperiosteal Implantation Injection
  Arms: Restylane® Perlane® Lidocaine

SUMMARY:
The cumulative effect of aging and environmental exposures (ie, ultraviolet, infrared, and visible light radiation and pollution) leads to wrinkles, discoloration, laxity, and roughness of sun exposed skin. The rapid restoration of soft tissue augmentation is commonly achieved by the use of dermal fillers. HArmonyCa Lidocaine injectable gel is a dermal filler intended for facial soft tissue augmentation. The purpose of this study is to assess adverse events and effectiveness of HArmonyCa Lidocaine injectable gel compared to Restylane® Perlane® Lidocaine (Perlane) in adults seeking restoration and/or correction of moderate to severe mid-face volume deficit.

HArmonyCa Lidocaine Injectable Gel is an investigational device being developed for soft tissue augmentation in the mid face. Participants are placed in 1 of 2 groups, called treatment arms. There is a 1 in 3 chance that participants will be assigned to the receive active comparator, Perlane. Around 252 adult participants seeking restoration and/or creation of mid-face volume will be enrolled in the study at approximately 9 sites in China.

Participants will receive HArmonyCa Lidocaine injectable gel or Perlane at Day 1 with an option touch-up treatment on Day 31. Participants will be followed for up to 12 Months after last treatment.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Has moderate (3), significant (4), or severe (5) mid-face volume deficit on the Mid-face Volume Deficit Scale (MFVDS) 5-point photonumeric scale based on evaluating investigator (EI) live assessment at randomization visit.
* Mid-face areas are amenable to achieving at least a 1-point improvement in MFVDS score with the allowed injection volume in the treating investigator's (TI) judgment.
* Must be in good health as determined by medical history, physical examination, vital signs, and investigator's judgment, including no known active pandemic infection.

Exclusion Criteria:

* Excessive skin laxity in the mid-face area in the opinion of the TI.
* Significant skin pigmentation disorders or discoloration in the mid-face area that would interfere with the visual assessment of the mid-face area.
* Semi-permanent soft tissue filler treatment (e.g., CaHA, poly-L-lactic acid) in the face within 36 months before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status Based on the Evaluating Investigator's (EI) Live Assessment of Mid-Face Volume Deficit Scale (MFVDS) | Month 6
  A "responder" is a participant with at least 1-point improvement (reduction) of mid face volume deficit using the MFVDS. MFVDS is a validated 5-point scale (1 = None/Minimal to 5 = Severe).
Number of Participants with Adverse Events (AEs) | Up to Approximately Month 14
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a medical device which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status Based on EI's Assessments of Global Aesthetic Improvement in the Treatment Area Using the Global Aesthetic Improvement Scale (GAIS) | Month 6
  A "responder" is a participant who achieves "Improved" or "Much Improved" on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the treatment area (2 = Much Improved, -2 = Much Worse).
Percentage of Participants Achieving "Responder" Status Based on Participant's Assessments of Global Aesthetic Improvement in the Treatment Area Using GAIS | Month 6
  A "responder" is a participant who achieves "Improved" or "Much Improved" on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the treatment area (2 = Much Improved to -2 = Much Worse).
Change from Baseline on the Overall Score of FACE-Q Satisfaction with Cheeks | Month 6
  The FACE-Q Satisfaction with Cheeks questionnaire is a 5-point survey where 1 = Very Dissatisfied and 4 = Very Satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (9):
- China (9):
  - Beijing Hospital /ID# 272476, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (West) - Xidan Campus /ID# 272480, Beijing, Beijing Municipality
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 272631, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 272468, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 272471, Nanjing, Jiangsu
  - Wuxi People'S Hospital /ID# 275928, Wuxi, Jiangsu
  - Huashan Hospital Of Fudan University /ID# 272632, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital /ID# 272509, Shanghai, Shanghai Municipality
  - The First People's Hospital of Hangzhou /ID# 272475, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-782